CLINICAL TRIAL: NCT04216056
Title: Evaluation of a Frailty Intervention Program in Hong Kong: A Pre-Post Study and a Focus Group Study
Brief Title: Evaluation of a Frailty Intervention Program in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jean Woo, Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019.455
Record Dates: First submitted 2019-12-23; First posted 2020-01-02 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frailty intervention program (Experimental): There will be 2 sessions per week for 12 weeks. Each session includes 1 hour exercise (including 5-10 minute warm-up and cool-down routine, 20-30 minute chair-based resistance exercises using Thera-Bands for muscle groups in both the upper and lower body, and 20-30 minutes aerobic exercises); and 1 hour game training using computer video games, board games and card games. Nutrition education will be given to the subjects based on their weight status. The 1st level of nutrition information (healthy eating tips for frailty prevention and management) will be given to all subjects on regular basis during the 12-week study period via short videos, text messages or Whatsapp reminders. On top of the 1st level nutrition information, 3 nutrition heath talks (1-1.5 hours per talk) about weight management will be given to those with BMI >=25 kg/m2, and/or waist circumference >=90 cm (male) or >=80 cm (female) during the 12-week study period.
  Interventions: Behavioral: Frailty intervention program
- Control group (No Intervention): Subjects in the control group will be asked to maintain their usual diet and physical activity patterns over the 12 weeks.

INTERVENTIONS:
Behavioral: Frailty intervention program — There will be 2 sessions per week for 12 weeks. Each session includes 1 hour exercise (including 5-10 minute warm-up and cool-down routine, 20-30 minute chair-based resistance exercises using Thera-Bands for muscle groups in both the upper and lower body, and 20-30 minutes aerobic exercises); and 1 hour game training using computer video games, board games and card games. Nutrition education will be given to the subjects based on their weight status. The 1st level of nutrition information (healthy eating tips for frailty prevention and management) will be given to all subjects on regular basis during the 12-week study period via short videos, text messages or Whatsapp reminders. On top of the 1st level nutrition information, 3 nutrition heath talks (1-1.5 hours per talk) about weight management will be given to those with BMI >=25 kg/m2, and/or waist circumference >=90 cm (male) or >=80 cm (female) during the 12-week study period.
  Arms: Frailty intervention program

SUMMARY:
The present study aims to compare the pre-post effect of a frailty intervention program with exercise, nutrition, cognitive and social components with a control group without such program on improving gait speed and frailty in community-dwelling Chinese adults aged 50 and above who are pre-frail or frail using the FRAIL scale, and to obtain their views towards the frailty intervention program. The investigators hypothesized that the frailty intervention program will result in improvements regarding frailty, mobility, weight status and other health outcomes.

This study will be a non-randomized controlled study using a controlled before-and-after study design. Eligible subjects will be assigned to one of the two groups: frailty intervention program, or control group without any intervention, over 12 weeks. A total of 152 subjects (76 per group) will be recruited. A sub-sample of 25 subjects from the intervention group will be invited to share their experience and opinion in focus groups.

DETAILED DESCRIPTION:
A 30-month trial, which will be divided into three phases, namely study preparation and subject recruitment (6 months), data collection (18 months), and data entry and analysis (6 months), will be conducted.

This study will be a non-randomized controlled study using a controlled before-and-after study design. Eligible subjects will receive a baseline assessment in the community facilities. After that, eligible subjects will be assigned to one of the two groups: frailty intervention program, or control group without any intervention, over 12 weeks. Subjects in the frailty intervention program will be invited to participate in the following components: exercise, game training and nutrition education; while subjects in the control group will be asked to maintain their usual diet and physical activity patterns. A total of 152 subjects (76 per group) will be recruited. Outcome measurements will be collected at two time points, namely baseline (T0), and 12 (T1) weeks.

The primary outcome will be the improvement in gait speed over 12 weeks. Secondary outcomes will include the change in the following parameters over 12 weeks: frailty, handgrip strength, 5 chair stands, balance test, Frontal Assessment Battery, dietary intake, nutritional status, physical activity, self-rated health, life satisfaction and self-efficacy of chronic disease management. In a sub-sample of 25 subjects from the intervention group, their views towards the frailty intervention program will be obtained from the focus group study.

ELIGIBILITY:
Inclusion Criteria:

* People aged 50 years or older;
* FRAIL score ≥ 1, and thus are considered pre-frail / frail;
* Chinese origin;
* Normally reside in Hong Kong;
* Could speak and understand Chinese;
* Willing to follow the study procedures.

Exclusion Criteria:

* Live in a residential aged care facility;
* Recent (i.e. past 3 months) or concurrent participation in any clinical trial or exercise and/or cognitive and/or dietary intervention program;
* With medical advice or conditions prohibiting exercise or medical conditions that precluded safe participation in an exercise program;
* With any other indication of a major medical or psychological illness, as judged by the investigators as ineligible to participate the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Change in gait speed | baseline, 12 weeks
  This outcome will be measured using the 6-meter walk test.

SECONDARY OUTCOMES:
Frailty status | baseline, 12 weeks
  Frailty status (i.e. robust, prefrail or frail) measured using the frailty scale (FRAIL) in which unabbreviated scale name is unavailable for this scale. Frailty scores from 0 to 5 (i.e., 1 point for each component; 0 = best to 5 = worst) and represent robust (0), pre-frail (1-2), and frail (3-5) health status.
Handgrip strength | baseline, 12 weeks
  Handgrip strength will be measured using a dynamometer.
5 chair stands | baseline, 12 weeks
  Muscle endurance in the lower extremities - Participant will be required to rise from a chair a total of 5 times, as quickly as they could, with arms across their chest. The amount of time required to complete all 5 repetitions will be recorded.
Balance test | baseline, 12 weeks
  Participant will be required to stand with different postures and maintain balance for 10 seconds each. The number of completed posture will be used for analysis.
Cognitive performance | baseline, 12 weeks
  Frontal Assessment Battery will be used to assess executive function. Total score is a maximum of 18, higher scores indicating better performance.
Dietary intake | baseline, 12 weeks
  Dietary habits and patterns over the past week will be assessed using a questionnaire designed by the research team based on the questionnaire used in the Hong Kong Child Health Survey (Department of Health, 2009) with modifications.
Nutritional status | baseline, 12 weeks
  This outcome will be assessed using Mini-Nutritional Assessment Short Form (MNA-SF). The total score of the MNA-SF ranges from 0-14 points, with 0-7 points indicate malnourished, 8-11 points as at risk of malnutrition and 12-14 points as normal nutritional status.
Physical activity | baseline, 12 weeks
  This outcome will be assessed using a validated Chinese version of the International Physical Activity Questionnaire (IPAQ-C). Metabolic equivalent for Task (MET)-minutes/week values for walking, moderate-intensity activities, vigorous-intensity activities, and total physical activities will be calculated for data analysis. Higher MET-minutes/week value represents higher amount of energy expended in carrying out physical activity.
Self-rated health | baseline, 12 weeks
  This outcome will be elicited by a single question, "Generally speaking, how is your health: excellent, very good, good, fair, or poor?" .
Life satisfaction | baseline, 12 weeks
  This outcome will be assessed by the subjects' response to the question "Are you satisfied with life?", using a 0 to 10-point linear scale. Higher point represents better self-rated life satisfaction.
Self-efficacy of chronic disease management | baseline, 12 weeks
  This outcome will be assessed using a validated Chinese version of short-form Chronic Disease Self-Efficacy Scales (CDSES) for older adults. Each item will be rated by the subjects on a scale from 1-10. The total score of the short-form CDSES is the mean of the six items, with higher score indicates better self-efficacy.
Views towards the frailty intervention program | 12 weeks
  Participants in the intervention group will be invited to share their experience and opinion in focus groups (of 1 to 1.5 hours duration).

OTHER OUTCOMES:
Weight | baseline, 12 weeks
  Weight in kilogram measured using standardized method.
Height | baseline, 12 weeks
  Height in centimeter measured using standardized method.
Waist circumference | baseline, 12 weeks
  Waist circumference in centimeter measured using standardized method.
Systolic blood pressure | baseline, 12 weeks
  Systolic blood pressure in mmHg measured using standardized method.
Diastolic blood pressure | baseline, 12 weeks
  Diastolic blood pressure in mmHg measured using standardized method.
Fat mass percentage | baseline, 12 weeks
  This outcome will be measured using bioelectrical impedance analysis (BIA).
Fat free mass percentage | baseline, 12 weeks
  This outcome will be measured using bioelectrical impedance analysis (BIA).

CONTACTS AND LOCATIONS:
Overall Officials: Jean Woo, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, China